CLINICAL TRIAL: NCT05772130
Title: Family HOPE Study (Hereditary Lynch Syndrome Opportunities for Participation &Amp; Engagement)
Brief Title: Provider-Mediated Communication of Genetic Testing Results to At-Risk Relatives of Cancer Patients to Improve Genetic Counseling and Testing Rates, Family HOPE Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22261; NCI-2023-01626 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22261 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Hereditary Malignant Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (usual care) (Active Comparator): Patients receive a family letter and their genomic test report to share with at-risk first degree relatives on study.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review; Other: Survey Administration
- Arm II (provider-mediated contact) (Experimental): Patients receive a family letter and their genomic test report to share with at-risk first degree relatives and relatives also receive provider-mediated contact to discuss genetic results on study.
  Interventions: Other: Electronic Health Record Review; Behavioral: Personal Contact; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive family letter and genomic test report
  Other Names: standard of care; standard therapy
  Arms: Arm I (usual care)
Other: Electronic Health Record Review — Ancillary studies
Behavioral: Personal Contact — Receive family letter and genomic test report with provider-mediated contact
  Other Names: Contact
  Arms: Arm II (provider-mediated contact)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial tests whether provider-mediated communication of genetic testing results to at-risk relatives of cancer patients can help improve genetic counseling and testing rates. Approximately 15% of people with cancer have an inherited form of cancer due to changes in a gene that they have inherited from one of their parents. These changes increase a person's risk for developing cancer. Most people who have an inherited harmful change in a cancer risk gene don't know that they have it and are therefore not able to get the health care that they need. The primary reason for this problem has been a lack of genetic counseling and testing for cancer patients and patients with a strong family history of cancer. Another reason for this lack of awareness is that, when cancer runs in a family, the patient who carries the gene change usually has to communicate the genetic risk information to their family members. When this process doesn't work well, family members may not know that they need to get genetic testing and then may not get potentially life-saving care. Provider-mediated contact to discuss genetic test results may help improve rates of genetic testing among at-risk relatives of patients with a family cancer syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Improve rates of family member cascade testing. II. Evaluate the psychosocial impact of provider-mediated contact to communicate genetic testing results.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Patients receive a family letter and their genomic test report to share with at-risk first degree relatives on study.

ARM II: Patients receive a family letter and their genomic test report to share with at-risk first degree relatives and relatives also receive provider-mediated contact to discuss genetic results on study.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Enrolled in City of Hope (COH) institutional review board (IRB) 07047 or have been seen by COH Genetics for genetic testing
* PATIENTS: Have an pathogenic/ likely pathogenic germline variant
* PATIENTS: Fluent in English
* PATIENTS: Age >= 18 years
* PATIENTS: Willing to provide contact information for eligible first-degree relatives
* PATIENTS: >= 2 first-degree relatives that are eligible for genetic testing and reside in the United States of America
* FIRST-DEGREE RELATIVES: Proband is a COH patient and has consented to this study
* FIRST-DEGREE RELATIVES: First-degree relative of proband
* FIRST-DEGREE RELATIVES: Resides within the United States
* FIRST-DEGREE RELATIVES: Has not undergone genetic testing for the known familial variant
* FIRST-DEGREE RELATIVES: Are fluent in English
* FIRST-DEGREE RELATIVES: Age >= 18 years

Exclusion Criteria:

* PATIENTS: Unable to provide informed consent
* PATIENTS: =< 2 at-risk first-degree relatives who are eligible for genetic testing and/or reside within the United States
* PATIENTS: Unwilling to provide contact information for family members
* FIRST-DEGREE RELATIVES: Unable or unwilling to provide informed consent
* FIRST-DEGREE RELATIVES: Have undergone genetic testing for the known familial variant
* FIRST-DEGREE RELATIVES: Resides outside of the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2026-12-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
The percentage of uptake of cascade testing among patients' first-degree at-risk relatives | Up to 9 months after enrollment
  Will calculate descriptive statistics first, including the mean, median and standard deviation of the number of the first-degree and secondary-degree at-risk relatives. We will then compare the proportion of identified relatives who completed genetic testing between the intervention and the control arms with a one-sided Cochran-Mantel-Haenszel test. Type I error of 0.05 will be used and descriptive statistics will be calculated for all exploratory outcomes along with 95% confidence intervals. All statistical testing and calculation of confidence intervals will adjust for intra-proband correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy W Gray, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States